CLINICAL TRIAL: NCT00004744
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Intravenous Immune Globulin for Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Mayo Clinic (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11660; MAYOC-27992
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immune globulin

SUMMARY:
OBJECTIVES: I. Determine whether high-dose intravenous immune globulin (IVIG) is more effective than placebo in restoring neurologic function (muscle strength) in patients with multiple sclerosis.

II. Determine the time to recovery following IVIG.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are treated with intravenous immune globulin or placebo. In the absence of a hypersensitivity reaction to a test dose, a total of 11 doses is administered: daily for 5 days, then every 2 weeks for 12 weeks.

Patients are followed at 3 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinically or laboratory-supported definite multiple sclerosis
* Disease relapsing-remitting or relapsing-progressive (i.e., secondary- progressive)
* Targeted neurologic deficit as follows: 25% or more loss of power in at least 1 limb Severity -1 or greater on Mayo Clinic rating scale OR Between 3+/5 and 4-/5 on Medical Research Clinic muscle power scale
* Documented by Mayo Clinic Department of Neurology as neither progressing nor improving for 4 to 18 months prior to entry No clinical evidence of spontaneous or corticosteroid-induced improvement
* Able to cooperate with isometric strength testing requirements

--Prior/Concurrent Therapy--

* No concurrent experimental drug therapy
* No concurrent intravenous immune globulin At least 3 months since immunosuppressive therapy, e.g., corticosteroids and corticotropin
* At least 3 months since plasma exchange

--Patient Characteristics--

* Hepatic: No coagulation defect, e.g., hyperviscosity syndrome
* Renal: Creatinine no greater than 1.5 times normal
* Cardiovascular: No unstable or advanced ischemic or cerebrovascular disease, e.g.: angina congestive heart failure transient ischemic attack stroke
* Immunologic: No human gamma globulin or albumin sensitivity No hypergammaglobulinemia No known antibody deficiency syndrome, especially IgA deficiency

Other:

* No condition interfering with neurologic exam, e.g.:
* Major amputation
* Deforming arthritis
* Major psychiatric illness
* Superimposed lower motor neuron deficit
* No intellectual impairment precluding study participation
* No pregnant or nursing women
* Adequate contraception required of fertile patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76
Dates: Start 1993-02; Primary Completion 1998-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Noseworthy, Study Chair — Mayo Clinic